CLINICAL TRIAL: NCT02599389
Title: Economic Evaluation Comparing Standard Balloon Angioplasty Versus Drug-eluted Balloon or Laser-Excimer in Association With Drug-eluted Balloon in the Treatment of Femoropopliteal Artery In-stent Restenosis.
Brief Title: Comparison of Angioplasty/Drug Coated Balloon/Laser + Drug Coated Balloon for Femoropopliteal Artery In-stent Restenosis
Acronym: INTACT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2014/40
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Angioplasty, Balloon
Keywords: in-stent restenosis; drug-coated balloons; Excimer Laser, cost effectiveness study, quality of life
MeSH Terms: interventions — Lasers, Excimer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard balloon (No Intervention): Angioplasty with use of standard balloons
- Drug-coated balloons (Experimental): Angioplasty with use of drug-coated balloons
  Interventions: Device: Drug-coated balloons
- Drug-coated balloons and laser (Experimental): Angioplasty with use of drug-coated balloons in association with Excimer Laser
  Interventions: Device: Drug-coated balloons; Device: Excimer Laser

INTERVENTIONS:
Device: Drug-coated balloons
  Other Names: In.Pact (Medtronic)
  Arms: Drug-coated balloons; Drug-coated balloons and laser
Device: Excimer Laser
  Other Names: SPECTRANETICS
  Arms: Drug-coated balloons and laser

SUMMARY:
The aim of this multicenter triple-arm randomized study is to compare two innovative techniques with the gold standard currently used and providing unsatisfactory results for the In-Stent Restenosis (ISR) treatment in femoro-popliteal arteries. This protocol compares the use of drug-coated balloons (paclitaxel - antimitotic) used alone or in association with the Excimer Laser to recalibrate the vessel lumen into the stent by destroying the whole fibrous material to the standard angioplasty using plain balloons. INTACT study main objective is to assess cost-effectiveness ratio of the treatment of femoropopliteal artery in-stent restenosis by comparing these two innovative strategies and the standard one in terms of cost per Qaly (Quality adjusted life-years) gained at 18 months from a collective perspective.

DETAILED DESCRIPTION:
The publication show that there is probably an effectiveness gradient (expressed as a proportion of patients with in-stent restenosis a 18 months after the intervention of the first stenosis reduction): standard balloons would be less effective than active balloons themselves less effective than in combination with the excimer laser. Reducing the risk of In-Stent Restenosis has major implications for the treatment of patients because it reduces the use of arterial bypass or amputation, if unable to perform revascularization.

Based on these promising results of efficiency, we can hypothesize that the active balloons in combination with the Excimer laser would improve the quality of life of patients while reducing the cost of their treatment, this compared to only assets balloons. This same improvement in quality of life with reduced costs of care would be observed for only assets compared to standard balloons. In health economic terms, it is therefore likely that the strategy combining assets balloons and Excimer laser is dominant over assets balloons themselves dominant over standard balloons.

ELIGIBILITY:
Inclusion Criteria:

* Patient of age > 18 years
* Patient with previously peripheral implanted stent(s) located in or extending to the popliteal artery
* Patient who received this stent between 3-36 months before inclusion
* Patient with one or more in-stent restenosis lesion(s) > 70% in the same arterial segment in association with clinical symptoms of claudication or an critical limb ischemia with Rutherford classification of 2, 3, 4 or 5
* Reference vessel diameter between 4 and 7 mm
* Patient affiliated to a social security regimen
* EC-approved consent form signed by the participant and the investigator (must be signed prior initiation of any study related intervention)

Exclusion Criteria:

* Life expectancy >18 months
* Patient already included in this study (recruitment of the contralateral leg is not allowed)
* Patient contraindicated for the use of antiplatelet therapy
* Pregnant or breast-feeding women
* Patient with a target limb infection being treated
* Patient with a procoagulant blood disease
* Patient with history of contrast agents allergies
* Patient with intolerance to paclitaxel
* Patient with severe renal impairment (GFR <30 ml / min / 1.73 m²) or patient with a creatinine clearance <15 ml / min
* External compression of previously implanted stent
* Patient participating in any clinical trial using another investigational drug or product which could interfere with the interpretation of the trial results.
* Patient under trusteeship or guardianship

Angiographic exclusion criteria :

* Inflow (above) severe lesion >70% or occlusion untreated satisfactorily (residual lesion> 50%) before the management of the target lesion
* Perforation, dissection or lesions on the arterial network access requiring an assumption prior to randomization
* Stent fracture grade 4 or 5 at the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Incremental cost per Qaly gained at 18 months | 18 months after angioplasty
Incremental cost per avoided stenosis relapse at 18 months | 18 months after angioplasty

SECONDARY OUTCOMES:
New In-stent restenosis during follow-up | 1 month, 6 months, 12 months and 18 months after angioplasty
  No recurrence of in-stent restenosis > 50% during follow-up with doppler . The three treatment groups are compared.
A major adverse event | 1 month, 6 months, 12 months and 18 months after angioplasty
  Absence of major event during follow-up as death, lower limb amputation or lack of required revascularization.
Improvement in the walking procedure | Before and 12 months after angioplasty
  Improvement in the walking procedure performing by Strandness test
Clinical improvement | 6 months, 12 months and 18 months after angioplasty
  Clinical improvement by the Rutherford classification at 6, 12 and 18 months. This improvement is objectified by a decrease in category 1 or several classes.
Systolic blood pressure Index | 6 months, 12 months and 18 months after angioplasty
  Index :ratio of brachial pressure and compressible leg artery pressure
new treatment for the treated lesion | 6 months, 12 months and 18 months after angioplasty
revascularization, with restenosis of the treated lesion | 6 months, 12 months and 18 months after angioplasty
recurrence of clinical symptoms | 6 months, 12 months and 18 months after angioplasty
Blood ultrasonic doppler velocimetry | 6 months, 12 months and 18 months after angioplasty

CONTACTS AND LOCATIONS:
Overall Officials: Eric DUCASSE, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — Unité de Soutien Méthodologique à la Recherche clinique et épidémiologique; University Hospital, Bordeaux
Locations (15):
- France (15):
  - Clinique Rhône Durance, Avignon
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - University Hospital of Bordeaux - Hospital Pellegrin, Bordeaux
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Hospices Civils de Lyon, Lyon
  - Hôpital Timone Adultes, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Polyclinique Les Fleurs, Ollioules
  - Hôpital Européen Georges Pompidou - AP-HP de Paris, Paris
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Clinique de L'Europe, Rouen
  - Centre Hospitalier Universitaire de St Etienne, Saint-Etienne
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
  - Clinique Pasteur, Toulouse